CLINICAL TRIAL: NCT05421312
Title: Periarticular Penetration of Cefazolin and Clindamycin in Second Stage Revision Arthroplasty of the Hip
Acronym: CONCENTRATE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-13583
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: PJI; Bone and Joint Infection; Pharmacokinetics
MeSH Terms: interventions — Cordocentesis

STUDY DESIGN:
Intervention Model Description: This explorative, low intervention study will be conducted in the Radboudumc Nijmegen and Sint Maartenskliniek (SMK) Nijmegen, The Netherlands.
  Subject will receive the cefazolin antibiotic prophylaxis and clindamycin antibiotic therapy as standard of care. The study interventions will include blood sampling on baseline and perioperative sampling of serum, synovial fluid and bone for the concentration measurements of the antibiotic agents. For every participating subject 3 serum samples, 1 synovial fluid sample and 2 bone samples will be taken for concentration measurement of cefazolin and clindamycin. Samples will be taken at different timepoints during the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cefazolin (Other): The cefazolin antimicrobial prophylaxis (2000mg single dose intravenously 15-60 minutes before incision) is part of standard of care.
  Interventions: Drug: sampling blood; Drug: Sampling synovial fluid; Drug: Sampling bone tissue
- Clindamycin (Other): The clindamycin (600mg three times daily orally) PJI therapy is part of standard care.
  Interventions: Drug: sampling blood; Drug: Sampling synovial fluid; Drug: Sampling bone tissue

INTERVENTIONS:
Drug: sampling blood — During the reimplantation, 3 serum samples will be taken at different timepoint during the procedure.
Drug: Sampling synovial fluid — During the reimplantation 1 synovial fluid sample will be taken prior to incision.
Drug: Sampling bone tissue — During the reimplantation 2 cortical bone samples will be taken at different timepoints during the procedure.

SUMMARY:
To prevent periprosthetic joint infection (PJI), optimal penetration of antibiotics into the joint-space is needed. In revision arthroplasty, the incidence of PJI is increased compared to primary arthroplasty. In this study, the penetration of antibiotic agents into the synovial fluid and bone will be analyzed. The concentration of antibiotics will be related tot the to the susceptibility (minimal inhibitory concentration; MIC-90) of microorganisms that frequently cause PJI.

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) is a feared complication of joint replacement, with an incidence of 0.5-1% after primary joint replacement and 3-5% after revision arthroplasty. For orthopaedic surgery involving a prosthesis, the administration of systemic antibiotic prophylaxis is strongly recommended to prevent PJI. Cefazolin is widely used as agent of choice in surgical antibiotic prophylaxis. Previous studies, all performed in patients undergoing primary joint replacement, demonstrated that the concentration of cefazolin in bone and synovial fluid was dose-dependent and exceeds the MIC90 for methicillin susceptible Staphylococcus aureus (MSSA), when given as 1 to 4 gram single dose shortly before incision. When a PJI is already present, clindamycin is used as treatment option in PJI caused by staphylococci (when combined with rifampicin) or cutibacteria. A limited number of studies have been performed to analyse the penetration of clindamycin into bone. These studies showed that clindamycin penetrates well into the bone and concentrations exceeded the MIC90 for MSSA. No studies have been performed to analyse the penetration of antibiotic agents into the periarticular tissue in patients who will undergo revision arthroplasty. In revision arthroplasty a foreign body (prosthesis) is in situ and periarticular tissue condition can be compromised due to previous surgical procedures and the presence of bone reaction to the prosthesis. It is not known whether the difference in PJI incidence after primary and revision arthroplasty may be explained by different penetration of the surgical antibiotic prophylaxis. The aim of this explorative study is to analyse the penetration of cefazolin and clindamycin into synovial fluid and bone and whether the concentration of the agents exceeds the MIC90 for micro-organisms frequently causing PJI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 years or older.
2. Scheduled second stage revision arthroplasty (reimplantation) of the hip prosthesis during clindamycin 600mg three times a day orally for PJI, started at least 3 days before reimplantation (steady state).

Exclusion Criteria:

1. Antibiotic prophylaxis other than cefazolin 2000mg i.v.
2. Cefazolin use within 4 days previous to the reimplantation, other than the single dose administration of surgical prophylaxis just before incision.
3. Clindamycin loaded bone cement in situ.
4. BMI more than 35 kg/m2.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
penetration cefazolin into synovial fluid | during surgical procedure prior to incision the synovial fluid sample will be taken
  The ratio (%) of the concentration of cefazolin in synovial fluid to serum.
penetration cefazolin into bone tissue | during surgical procedure prior to incision the synovial fluid sample will be taken
  The ratio (%) of the concentration of cefazolin in synovial fluid to serum.
penetration clindamycin into bone tissue | during surgical procedure, directly after opening the joint and before reimplantation of the prosthesis the bone samples will be taken
  The ratio (%) of the concentration of cefazolin in bone tissue to serum.

SECONDARY OUTCOMES:
AUC/MIC90 of cefazolin | sampling during procedure
  The ratio of area under the curve of cefazolin to the minimal inhibitory concentration-90 of microorganisms
AUC/MIC90 of clindamycin | sampling during procedure
  The ratio of area under the curve of cefazolin to the minimal inhibitory concentration-90 of microorganisms
factors associated with reduced cefazolin concentration | sampling during procedure
  univariable and multivariable (if possible) analysis for factors that are associated with reduced concentration of cefazolin (i.e., BMI, age, ..)
factors associated with reduced clindamycin concentration | sampling during procedure
  univariable and multivariable (if possible) analysis for factors that are associated with reduced concentration of cefazolin (i.e., BMI, age, ..)

CONTACTS AND LOCATIONS:
Overall Officials: Nynke Jager, PhD, Principal Investigator — Radboud University Medical Center; Jon Goosen, MD, PhD, Principal Investigator — Sint Maartenskliniek

IPD SHARING:
Plan to Share IPD: No